CLINICAL TRIAL: NCT07345260
Title: The Effects of a Nutritional Supplement on Sleep Quality
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Athletic Greens International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AG-20801
Record Dates: First submitted 2025-12-22; First posted 2026-01-15 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-12

CONDITIONS: Sleep; Sleep Quality
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Maltodextrin + Flavoring
  Interventions: Dietary Supplement: Placebo
- Novel Sleep Supplement (Experimental): Novel powdered sleep supplement
  Interventions: Dietary Supplement: Novel powdered sleep supplement

INTERVENTIONS:
Dietary Supplement: Novel powdered sleep supplement — A dietary sleep supplement consisting of vitamins, minerals, adaptogens, and whole food ingredients
  Arms: Novel Sleep Supplement
Dietary Supplement: Placebo — maltodextrin placebo
  Arms: Placebo

SUMMARY:
This study is a randomized, double-blind, placebo-controlled study of N=140 adult men and women with sub-clinical sleep issues. This study to assess the effect of a novel dietary supplement on sleep related outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Be male or female
2. Be aged 35-65.
3. Body Mass Index: ≥18.5 and ≤29.9 kg/m2
4. Anyone currently experiencing issues with falling asleep, staying asleep, or waking up during the night
5. Score of 7 or less on the RU-SATED validated sleep questionnaire.
6. Anyone willing to follow the study protocol.
7. Anyone willing to discontinue any other supplements (nootroptics, adaptogens, calming herbs), medications, herbal remedies, over the counter sleep medications [e.g., zolipidem, diphenhydramine (Benadryl or unisom), magnesium or melatonin products] used to assist with sleep for the duration of the study.
8. Agree to limit alcohol intake within ~4 hours of bedtime
9. Agree to limit caffeine intake to ≤ 400 mg/day (~3-4 cups of coffee) or ingestion of caffeine-containing products after 2:00 PM during the study period.
10. Anyone who is generally healthy - does not live with any uncontrolled chronic disease.
11. Resides in the United States.

Exclusion Criteria:

1. Anyone with a diagnosed chronic sleep condition, including but not limited to insomnia, narcolepsy, REM Behavior Disorder, moderate to severe restless leg syndrome (RLS), or sleep apnea.
2. Women currently undergoing perimenopause or experiencing vasomotor symptoms such as night sweats.
3. Use of hormone therapy (including estrogen, progesterone, or phytoestrogens) within the last 3 months.
4. Anyone with diagnosed psychiatric disorders including major depressive disorder with acute symptoms, Bipolar disorder, Generalized anxiety disorder with active symptoms, PTSD with frequent nightmares
5. Anyone with diagnosed neurogenitive diseases or chronic pain disorders including Parkinson's disease, Alzheimer's disease, or uncontrolled fibromyalgia
6. Anyone who regularly consumes prescribed stimulant medications including Amphetamines (e.g., Adderall, Vyvanse), Methylphenidate (e.g., Ritalin, Concerta), and Modafinil / Armodafinil
7. Anyone currently on CNS activating anti-depressants including Bupropion (Wellbutrin), Fluoxetine, Venlafaxine (Effexor), Sertraline (Zoloft).
8. Current or recent use of cannabis or THC-containing products, including recreational or medicinal marijuana, CBD products with measurable THC content, or synthetic cannabinoids, within the past 30 days.
9. Anyone with a job that disrupts their nighttime sleep (e.g., excessive travel, night/3rd shift workers).
10. Anyone unwilling to wear the Oura ring device for the duration of the trial or unwilling to open the Oura application at least three times each week during the trial for data to sync to the cloud
11. Anyone currently taking a prescription sleep aid.
12. Anyone who introduces any new supplements, medications, herbal remedies, or melatonin products used to assist with sleep for the duration of the study.
13. Anyone with any allergies or sensitivities to any of the study product ingredients.
14. Any women who are pregnant, breastfeeding, or trying to conceive (or who will be at any point during the study period).
15. Anyone with a history of substance abuse.
16. Anyone who drinks heavily (i.e., 8 or more alcoholic drinks per week for women or 15 or more alcoholic drinks per week for men).
17. Currently partaking in another research study or will be partaking in any other research study for the next 7 weeks, or at any point during this study's duration.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2026-01-02 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Tracked sleep activity | 42 days
  Assessed via Oura ring
Sleep quality | Baseline, week 3, and week 6
  Pittsburgh Sleep Quality Index and Restorative Sleep Questionnaire weekly

SECONDARY OUTCOMES:
Dietary habits | Baseline and endpoint (week 6)
  Automated Self-Administered 24-Hour (ASA24®) Dietary Assessment Tool
Oura Actigraphy - Daytime Activity | 42 days
  Daytime activity

OTHER OUTCOMES:
Comprehensive Metabolic Blood Panel | Baseline and endpoint (week 6)
  Serum concentrations of sodium, potassium, carbon dioxide, chloride, albumin, total protein, glucose, and calcium, ALT, AST, bilirubin, BUN, creatinine
Complete blood count | Baseline and endpoint (week 6)
  Circulating concentrations of white blood cells, red blood cells, hemoglobin, and hematocrit

CONTACTS AND LOCATIONS:
Overall Officials: Ellen O'Gorman, Principal Investigator — Citruslabs
Locations (1):
- Citruslabs, Santa Monica, California, United States